CLINICAL TRIAL: NCT07010003
Title: Ear Acupressure for Reducing Anxiety and Pain During Heart Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Robert Bosch-Krankenhaus Stuttgart (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 643/2024BO1
Record Dates: First submitted 2025-05-09; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Elective Heart Surgery
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): Standard preoperative care
- NADA-Acupressure (Experimental): Participants in the intervention arm of the study receive standardized ear acupressure treatment according to the NADA protocol before surgery.
  Interventions: Procedure: Acupressure

INTERVENTIONS:
Procedure: Acupressure — Ear acupressure following the NADA Protocol is carried out using special acupuncture patches that press a small bead onto defined points on the ear: Shen Men, kidney, lung, liver, and vegetative. NADA ear acupressure is a non-invasive and low-risk intervention. In addition, the protocol is carried out exclusively by NADA-certified doctors, medical assistants, or nursing staff.
  Arms: NADA-Acupressure

SUMMARY:
Acupuncture and acupressure, rooted in Traditional Chinese Medicine, are used to treat a variety of symptoms. One specific and easy-to-apply method is ear acupuncture/acupressure following the NADA protocol (developed by the National Acupuncture Detoxification Association in 1985 in New York). This technique has been used successfully in Germany since 1995. It is known for its balancing and stabilizing effects on both body and mind, helping to reduce symptoms such as anxiety and stress, and promoting relaxation and inner calm.

Open-heart surgery can be emotionally overwhelming for patients, often triggering intense existential fears. Preoperative anxiety may worsen physical and psychological symptoms and negatively affect surgery outcomes. Therefore, non-pharmacological interventions like acupuncture are gaining importance alongside medication.

Several studies have demonstrated the effectiveness of preoperative acupuncture in reducing pain, anxiety, and nausea across various surgeries. Randomized trials show significant anxiety reduction through both body and ear acupuncture. One study found that ear acupuncture can rapidly improve psychological well-being, with effects noticeable within five minutes. This suggests its potential use not only the day before surgery but also immediately beforehand.

In contrast, research on ear acupressure before heart surgery is limited. However, one study reported improvements in sleep quality and reduced anxiety. A recent review highlighted the positive effects of ear stimulation on stress, blood pressure, and heart rate, and even suggested that acupressure may be more effective than acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who are capable of giving consent or willing to do so and who are undergoing elective heart surgery at the Robert Bosch Krankenhaus study center are included.

Exclusion Criteria:

* Under 18 years old
* Emergency or urgent surgery
* Patients who are incapable of giving consent or unwilling to do so
* Patients who have received acupuncture treatment (including NADA ear acupuncture or acupressure) in the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Preoperative (Day 1)
  State-Trait Anxiety Inventory - state (STAI-s) The range of possible scores varies from a minimum of 20 to a maximum of 80, where higher scores represent higher anxiety.

SECONDARY OUTCOMES:
Anxiety | Baseline (Day 0, preoperative), Immediately after the acupressure session (Day 0, preoperative), Postoperative (Day 2 - Day 10 daily until discharged from hospital, on average 10 days)
  State-Trait Anxiety Inventory - state (STAI-s) The range of possible scores varies from a minimum of 20 to a maximum of 80, where higher scores represent higher anxiety.
Specific preoperative anxiety | Baseline (Day 0, preoperative), Immediately after the acupressure session (Day 0, preoperative), Preoperative (Day 1)
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) For the anxiety subscale, scores range between 4 and 20, higher scores reflect higher anxiety.
  For the need for information subscale, scores range between 2 and 10, higher scores reflect higher need for information
Quality of life | Baseline (Day 0, preoperative), Discharge from hospital (Day 10 on average)
  EQ5D
Pain intensity | Baseline (Day 0, preoperative), Postoperative (Day 2 - Day 10 daily until discharged from hospital
  Numerical Rating Scale Scores range between 0 and 10, higher scores indicate higher pain intensity
Depression | baseline (Day 0, preoperative)
  Beck Depression Inventory (BDI) Scores range between 0 and 63, with higher scores representing more severe depression symptoms.
Postoperative Nausea and Vomiting | Postoperative (Day 2)
  PONV
Major Adverse Cardiac and Cerebrovascular Events | Discharge from hospital (Day 10 on average)
  MACCE

CONTACTS AND LOCATIONS:
Overall Officials: Nora Göbel, Dr. med., Principal Investigator — Robert Bosch Medical Center
Locations (1):
- Robert Bosch Krankenhaus, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No